CLINICAL TRIAL: NCT03417349
Title: Safety and Effectiveness of SOFIA™/SOFIA™ PLUS When Used for Direct Aspiration as a First Line Treatment Technique in Patients Suffering an Acute Ischemic Stroke in the Anterior Circulation
Brief Title: Safety and Effectiveness of SOFIA™/SOFIA™ PLUS for Direct Aspiration in Acute Ischemic Stroke
Acronym: SESAME
Status: Completed | Type: Observational
Sponsor: Dr. Markus Alfred Möhlenbruch (Other)
Collaborators: Microvention-Terumo, Inc. (Industry); Eppdata Hamburg (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Markus Alfred Möhlenbruch, Principle Investigator, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Other Study IDs: SESAME
Record Dates: First submitted 2018-01-16; First posted 2018-01-31 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Cerebrovascular Stroke; Stroke, Acute; Cerebral Stroke
Keywords: Acute Ischemic Stroke; Thrombectomy; Aspiration Thrombectomy; Observational study
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Aspiration thrombectomy: Patients with acute ischemic stroke of the anterior circulation whom the treating physician deemed eligible to be treated with SOFIA™/ SOFIA™ as a first line treatment technique
  Interventions: Device: Sofia

INTERVENTIONS:
Device: Sofia — The SOFIA™/ SOFIA™ PLUS Catheter will be used in removal/aspiration of emboli and thrombi following the CE marked Instructions For Use. Enrollment into the study does not change the routine care at the site provided to the patient requiring mechanical thrombectomy treatment.
  Other Names: Microvention - SOFIA Catheter; Microvention - SOFIA Plus Catheter

SUMMARY:
Sesame is a European, multi-center, single arm, prospective, observational registry.

Sesame aims to demonstrate that use of SOFIA™/SOFIA™ PLUS catheter for direct aspiration as a first line treatment technique is fast, safe and effective in patients suffering an Acute Ischemic Stroke when assessed at 24 hours, discharge and 90 days after treatment. 250 patients will be enrolled. All patients will be followed for 90 days or until death.

DETAILED DESCRIPTION:
Several publications describing the use of aspiration as a first line treatment technique in AIS patients have shown superior technical results with similar clinical outcomes to those seen when using a traditional stent retriever. They have also shown decreased procedure time and cost. The aim of this study is to show similar results in terms of speed, Effectiveness and safety when SOFIA™/ SOFIA™ PLUS is the catheter used for first line aspiration thrombectomy.

The SOFIA™ (Soft Torqueable Catheter Optimized For Intracranial Access) and SOFIA™ PLUS Catheter are single lumen, flexible catheters, designed with coil and braid reinforcement. The SOFIA™ / SOFIA™ PLUS catheters have a soft distal tip for easy navigation in tortuous vessels. The tip is steam shapable and the proximal shaft torquable to help steer around challenging bifurcations. The coil and braid construction provides enhanced kink resistance and 1:1 push / pull control. Once navigated to the site of the occlusion, the SOFIA™ / SOFIA™ PLUS catheters can be used in conjunction with an aspiration source, such as a pump or syringe, to facilitate aspiration thrombectomy of the occluded vessel. The SOFIA™ / SOFIA™ PLUS catheters have large lumens, developed to maximize aspiration power and capture of thrombus.

SESAME is a multi-center, single arm, prospective, observational registry of the SOFIA™/ SOFIA™ PLUS Catheter in Europe. Consecutive patients presenting within 6 hours of symptom onset with an anterior circulation large vessel occlusion (LVO) acute ischemic stroke (within the internal carotid artery and internal carotid terminus, middle cerebral -M1/M2 segments) will be treated using aspiration thrombectomy as first intention and site routine practice. Devices received CE-mark and will be used according to the 'Instructions For Use'.

The follow-up visits will occur at 24 +/- 12 hours, at patient discharge, and 90+/-14 days post-procedure.

Furthermore the study design is adaptive, prospectively stating interim analyses with specified stopping rules, which allow for the possibility of the study to terminate early based on either a determination of study success or of the futility to continue further enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 18
2. Demonstrated occlusion of the distal intracranial carotid artery, middle cerebral artery (M1 or M2) or anterior cerebral artery (A1 or A2) proven by CT and/or MRI
3. NIHSS ≥ 2 and ≤ 30 at screening
4. Start of the thrombectomy procedure within 6 hours of the onset of stroke symptoms
5. Pre event mRS ≤1
6. Patient or patient's legally authorized representative has received information about data collection and has signed and dated an Informed Consent Form

Exclusion Criteria:

1. Patient is more than 6 hours from symptom onset
2. Rapidly improving neurologic examination
3. Evidence of cerebral ischemia in the posterior circulation
4. Severe unilateral or bilateral carotid artery stenosis requiring stent treatment
5. Presence of an existing or pre-existing large territory infarction
6. Absent femoral pulses
7. Excessive vascular tortuosity that will likely result in unstable access
8. Pregnancy; if a woman is of child-bearing potential a urine or serum beta HCG test is positive
9. Known contrast product allergy
10. Patient has a severe or fatal comorbidity that will likely prevent improvement or follow up or that will render the procedure unlikely to benefit the patient
11. Evidence of intracranial hemorrhage (SAH, ICH, etc.)

Imaging exclusion criteria:

* Significant mass effect with midline shift or intracranial tumor
* Baseline non-contrast CT or DWI MRI evidence of a moderate/large core defined as extensive early ischemic changes of Alberta Stroke Program Early CT score (ASPECTS) 0-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 18 years of age presenting with an acute ischemic event in the anterior cerebral circulation that can be treated within 6 hours from AIS symptom onset. Those eligible to be treated with SOFIA™/ SOFIA™ PLUS will be enrolled after having signed an informed consent form (or having one signed on his or her behalf by a legally authorized representative).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical outcome | 90 days
  Dichotomization of patients into good functional outcome defined as a modified Rankin Score (mRS) ≤ 2 and bad functional outcome defined as mRS >2

SECONDARY OUTCOMES:
Safety - neurological | Prior to discharge / approximated 3-7 days
  Occurrence of major neurological events (stroke, intracranial hemorrhage, intracerebral hemorrhage, etc.)
Safety - procedural | 90 days
  Devices and procedure related adverse events within 90 days of follow up
ENT | Intra-procedure
  Infarct in a New Territory After Treatment Administration as seen on final control angiogram at the end of the procedure
sICH | 24 hours
  Occurrence of symptomatic intracranial hemorrhage (sICH) within 24 hours
Vessel damage | Intra-procedure
  Occurrence of intracranial vessel damage at the end of the procedure as seen on final control angiogram at the end of the procedure
Recanalization - Aspiration | Intra-procedure
  Proportion of patients having complete recanalization (TICI≥ 2b) just after first line aspiration treatment as seen on control angiogram
Recanalization - Other | Intra-procedure
  Proportion of patients having complete recanalization (TICI ≥ 2b) af-ter thrombectomy using an additional devices as seen on control angiogram
Time to recanalization- Aspiration | Intra-procedure
  Time from groin puncture to complete recanalization (TICI ≥ 2b) in patients after first line aspiration treatment as seen on control angiogram
Time to recanalization- Other | Intra-procedure
  Time from groin puncture to complete recanalization (TICI ≥ 2b) in patients after thrombectomy using an additional device as seen on control angiogram
Time to angio | Intra-procedure
  Time from CT-scan/MRI at the institution to groin access
Symptom onset | Pre-procedure
  Time from symptom onset to CT-scan/MRI
Neurological outcome 24 | 24 hours
  National Institutes of Health Stroke Scale (NIHSS) score at 24 hours, total and subscale scores
Neurological outcome discharge | Discharge / approximately 3-7 days
  National Institutes of Health Stroke Scale (NIHSS) score at discharge, total and subscale scores
Neurological outcome 90 days | 90 days / +/- 14 days
  National Institutes of Health Stroke Scale (NIHSS) score at 90 days, total and subscale scores
Degree of disability - discharge | Discharge/ approximately 3-7 days
  modified Rankin Score at discharge, total score
Degree of disability - 90d | 90 days / +/- 14 days
  modified Rankin Score at 90 day follow-up, total score
Quality of Life at 90 days | 90 days / +/- 14 days
  Quality of Life at 90 days assessed via PROMIS Scale v1.2 - Global Health, total score
Imaging | 24 hours
  Difference of Alberta stroke program early CT score (ASPECTs) scores in CT/MRI pretreatment vs. 24h, total scores
Imaging - perfusion | 24 hours
  In the subgroup of patients with additional perfusion CT (as per local standard of care): volume of saved brain tissue determined by predictive modeling
Health Economics -device | Intra-procedure
  Device costs (standardized cost of all devices as well as human resources and medication used during index procedure)
Health Economics - hospital | Discharge / approximately 3-7 days
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Möhlenbruch, MD, Principal Investigator — University Hospital Heidelberg
Locations (15):
- Austria (2):
  - Kepler Universitätsklinikum, Linz
  - Salzburger Landeskliniken, Salzburg
- France (5):
  - Le Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Groupe Hospitalier Universitaire Pitié Salpêtrière, Paris
  - Kremin Bicêtre- Paris Sud University, Paris
  - CHU de Toulouse Hôpital Purpan, Toulouse
- Germany (6):
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Schleswig-Holstein, Kiel
- Policlinico "G. Martino" di Messina, Messina, Italy
- Universitair Medisch Centrum Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided